CLINICAL TRIAL: NCT03219957
Title: A Phase I Study Assessing Single and Multiple Doses of AT-527 in Healthy and HCV-Infected Subjects
Brief Title: Study of AT-527 in Healthy and HCV-Infected Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atea Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: AT-01B-001
Record Dates: First submitted 2017-07-13; First posted 2017-07-18 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Chronic Hepatitis C; Hepatitis C; Hepatitis C, Chronic
Keywords: HCV; Hepatitis C Virus; RNA Viruses; Flavivirus; Liver Diseases; Hepatitis, Viral, Human; Flaviviridae Infections
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C; Liver Diseases; Hepatitis, Viral, Human; Flaviviridae Infections | interventions — AT-511

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AT-527 (Experimental)
  Interventions: Drug: AT-527
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo Comparator

INTERVENTIONS:
Drug: AT-527 — Ascending doses of AT-527 administered orally.
  Arms: AT-527
Other: Placebo Comparator — Matching placebo
  Arms: Placebo

SUMMARY:
This study has multiple parts. It will assess the safety, tolerability and pharmacokinetics (PK) of AT-527 in healthy subjects and subjects infected with hepatitis C virus (HCV). In addition, the study will assess the antiviral activity of AT-527 in subjects infected with HCV.

ELIGIBILITY:
Inclusion Criteria:

All subjects (healthy and HCV-infected subjects):

* Must agree to use two methods of birth control from Screening through 90 days after administration of the last dose of study drug
* Must have a negative pregnancy test at Screening and prior to dosing
* Minimum body weight of 50 kg
* Willing to comply with the study requirements and to provide written informed consent

Additional inclusion criteria for HCV-infected subjects:

* Must have not received prior treatment for HCV infection
* Documented clinical history compatible with chronic HCV infection
* Plasma HCV RNA ≥ 5.0 log10 IU/mL at Screening.

Exclusion Criteria:

All subjects (healthy and HCV-infected subjects):

* Pregnant or breastfeeding
* Infected with hepatitis B virus or HIV
* Abuse of alcohol or drugs
* Use of other investigational drugs within 28 days of dosing
* Other clinically significant medical conditions or laboratory abnormalities

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2017-07-06 (Actual); Primary Completion 2018-06-20 (Actual); Study Completion 2018-06-20 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Through Day 6 for subjects receiving a single dose
  Number of subjects experiencing treatment-emergent adverse events
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Through Day 35 for subjects receiving multiple doses.
  Number of subjects experiencing treatment-emergent adverse events

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of AT-527 | Day 1 for subjects receiving a single dose; Days 1 and 7 for subjects receiving multiple doses
  Maximum plasma concentration (Cmax)
Pharmacokinetics (PK) of AT-527 | Day 1 for subjects receiving a single dose; Days 1 and 7 for subjects receiving multiple doses
  Area under the concentration-time curve (AUC)
Antiviral Activity of AT-527 | Through Day 6 for subjects receiving a single dose; Through Day 35 for subjects receiving multiple doses.
  Change from baseline in plasma HCV RNA

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Jian Zhou, PhD, Study Director — Atea Pharmaceuticals, Inc.
Locations (2):
- Clinical Trial Site, Antwerp, Belgium
- Clinical Trial Site, Chisinau, Moldova

REFERENCES:
- [Result] Berliba E, Bogus M, Vanhoutte F, Berghmans PJ, Good SS, Moussa A, Pietropaolo K, Murphy RL, Zhou XJ, Sommadossi JP. Safety, pharmacokinetics and antiviral activity of AT-527, a novel purine nucleotide prodrug, in HCV-infected subjects with and without cirrhosis. Antimicrob Agents Chemother. 2019 Sep 9;63(12):e01201-19. doi: 10.1128/AAC.01201-19. Epub 2019 Sep 30. PMID 31570394